CLINICAL TRIAL: NCT06136156
Title: Measuring Vital Signs and Biomarkers From Mobile Device Videos
Brief Title: Video Vitals and Biomarkers
Status: Completed | Type: Observational
Sponsor: Maiv Health Inc. (Industry)
Responsible Party: Principal Investigator, Sandro Luna, Principal Investigator, Maiv Health Inc.
Other Study IDs: AX8
Record Dates: First submitted 2023-10-17; First posted 2023-11-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cardiometabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

SUMMARY:
The investigators are doing this research to study the ability of mobile devices to measure vital signs and biomarkers from video as compared to standard-of-care clinical office tools.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to stay in a seated position for 30 minutes
* Must be able to participate in a venous blood draw

Exclusion Criteria:

* Condition that prevents prolonged seated position
* Condition that restricts ability to provide venous blood sample

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults greater than 18 years old may participate in this research study
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Heart rate in beats per minute | 2 minutes
Blood pressure (systolic/diastolic) in millimeters of mercury (mmHg) | 2 minutes
Respiration rate in breaths per minute | 2 minutes
Oxygen saturation in SpO2 percentage | 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Luna, MD, Principal Investigator — Maiv Health Inc.
Locations (1):
- ARCpoint Labs of Cedar Park, Cedar Park, Texas, United States

IPD SHARING:
Plan to Share IPD: No